CLINICAL TRIAL: NCT03023020
Title: Management of High Bleeding Risk Patients Post Bioresorbable Polymer Coated Stent Implantation With an Abbreviated Versus Prolonged DAPT Regimen
Acronym: MASTER DAPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ECRI bv (Industry)
Collaborators: Cardialysis B.V. (Industry); European Cardiovascular Research Center (Network); University of Bern (Other); Terumo Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECRI-009
Record Dates: First submitted 2016-12-29; First posted 2017-01-18 (Estimated); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: High Bleeding Risk; Coronary Artery Disease; PCI
Keywords: Dual Antiplatelet Therapy
MeSH Terms: conditions — Coronary Artery Disease | interventions — Aspirin; Platelet Aggregation Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abbreviated antiplatelet regimen (Other): Dual antiplatelet therapy is discontinued immediately after randomization (i.e. 1 month post stent implantation), and a single antiplatelet agent is continued until at least 11 months post randomization (i.e. 12 months post stent implantation).
  In patients on oral anticoagulants, dual antiplatelet therapy is discontinued immediately after randomization (i.e. 1 month post stent implantation), and either Aspirin or Clopidogrel is continued until 5 months post randomization (i.e. 6 months post stent implantation). Oral anticoagulation is continued until at least 11 months post randomization (i.e. 12 months post stent implantation)
  Interventions: Drug: Aspirin; Drug: P2Y12 inhibitor
- Prolonged antiplatelet regimen (Other): Aspirin is continued for at least 11 months post randomization (i.e. 12 months post stent implantation), the P2Y12 inhibitor being taken at the time of randomization is continued for at least 5 months and up to 11 months post randomization (i.e. 12 months post stent implantation).
  In patients on oral anticoagulants, aspirin and Clopidogrel are continued for at least 2 months post randomization (i.e. 3 months post stent implantation) and up to 11 months post randomization (i.e. 12 months after stent implantation). Either aspirin or Clopidogrel is continued up to 11 months post randomization (i.e. 12 months post stent implantation)
  Interventions: Drug: Aspirin; Drug: P2Y12 inhibitor

INTERVENTIONS:
Drug: Aspirin — Dosing per current guidelines and local practice
  Other Names: antiplatelet agent
Drug: P2Y12 inhibitor — Dosing per current guidelines and local practice
  Other Names: antiplatelet agent

SUMMARY:
The study compares two lengths of medication therapy (a shortened versus a prolonged dual antiplatelet therapy) in order to prevent thrombus (blood cloth) formation after the successfully treatment for coronary heart disease with a drug covered stent (metallic tube).

This comparison will be done in patients who, compared to the average patient, are more likely to suffer from complications on antiplatelet therapy (bleeding). Both durations are within the current medical recommendations. The aim of this study is to help improve further standard antiplatelet duration guidelines.

DETAILED DESCRIPTION:
The study objective is to determine in a high bleeding risk patient population undergoing PCI under standardized treatment (within current guidelines and instructions for use and including the bioresorbable polymer coated Ultimaster sirolimus-eluting stent), whether abbreviated DAPT is non-inferior to prolonged DAPT regimen in terms of NACE within 12 months, whether abbreviated DAPT is non-inferior to prolonged DAPT regimen in terms of MACCE within 12 months and whether abbreviated DAPT is superior to prolonged DAPT regimen in terms of MCB within 12 months.

There are two treatment strategies:

* abbreviated dual anti-platelet therapy: dual antiplatelet therapy is discontinued and a single antiplatelet agent is continued until at least 11 months post randomization (i.e. 12 months post stent implantation). In patients on oral anticoagulants, dual antiplatelet therapy is discontinued and either Aspirin or Clopidogrel is continued until 5 months post randomization (i.e. 6 months post stent implantation). Oral anticoagulation is continued until at least 11 months post randomization (i.e. 12 months post stent implantation) OR
* prolonged dual anti-platelet therapy: aspirin is continued for at least 11 months post randomization (i.e. 12 months post stent implantation), the P2Y12 inhibitor being taken at the time of randomization is continued for at least 5 months and up to 11 months post randomization (i.e. 12 months post stent implantation). In patients on oral anticoagulants, aspirin and Clopidogrel are continued for at least 2 months post randomization (i.e. 3 months post stent implantation) and up to 11 months post randomization (i.e. 12 months after stent implantation). Therefore either aspirin or Clopidogrel is continued up to 11 months post randomization (i.e. 12 months post stent implantation)

The study design is an investigator-initiated, randomized, multi-center, clinical trial to be conducted in approximately 100 interventional cardiology centers in across the globe excluding USA. The study includes 2 x 2150 patients (i.e. 4300 patients) Randomization will occur at one month after the PCI procedure. The expected duration of participation for each patient is 14 months.

ELIGIBILITY:
Inclusion Criteria:

After index PCI, patients aged 18 years or more are eligible for inclusion into the study if the following criteria are met.

1. At least one among the HBR criteria (as defined below) is met.
2. All lesions are successfully treated with Ultimaster stent in the context of routine clinical care, i.e. post-procedural angiographic diameter stenosis <20% by visual estimation
3. Free from any flow-limiting angiographic complications (i.e. significant untreated dissection or major side-branch occlusion), which require prolonged DAPT duration based on operator's opinion.
4. All stages of PCI are complete (if any) and no further PCI is planned.

At randomization visit (one month after index PCI), the following criteria must be met:

1. Fulfilment of at least one HBR criterion (as defined below), or on the basis of post-PCI actionable (i.e. requiring medical attention) non-access site related bleeding episode
2. Uneventful 30-day clinical course, i.e. free from spontaneous MI, symptomatic restenosis, stent thrombosis, stroke and any revascularization (coronary and non-coronary) requiring prolonged DAPT
3. If not on OAC,

   1. Patient is on a DAPT regimen of aspirin and a P2Y12 inhibitor
   2. Patient with one type of P2Y12 inhibitor for at least 7 days (i.e. no switching between oral P2Y12 inhibitors has occurred in the previous 7 days)
4. If on OAC

   1. Patient is on the same type of OAC (e.g. Vitamin K antagonist or NOAC) for at least 7 days
   2. Patient is on clopidogrel for at least 7 days

Definition of HBR

Post-PCI patients are at HBR if at least one of the following criteria applies:

* Clinical indication for treatment with oral anticoagulants (OAC) for at least 12 months
* Recent (<12 months) non-access site bleeding episode(s), which required medical attention (i.e. actionable bleeding).
* Previous bleeding episode(s) which required hospitalization if the underlying cause has not been definitively treated (i.e. surgical removal of the bleeding source)
* Age equal or greater than 75 years
* Systemic conditions associated with an increased bleeding risk (e.g. haematological disorders, including a history of or current thrombocytopaenia defined as a platelet count <100,000/mm3 (<100 x 109/L), or any known coagulation disorder associated with increased bleeding risk.
* Documented anaemia defined as repeated haemoglobin levels <11 g/dl or transfusion within 4 weeks before randomization.
* Need for chronic treatment with steroids or non-steroidal anti-inflammatory drugs
* Diagnosed malignancy (other than skin) considered at high bleeding risk including gastro-intestinal, genito-urethral/renal and pulmonary.
* Stroke at any time or TIA in the previous 6 months
* PRECISE DAPT score of 25 or greater

Exclusion Criteria:

1. Treated with stents other than Ultimaster stent within 6 months prior to index procedure
2. Treated for in-stent restenosis or stent thrombosis at index PCI or within 6 months before
3. Treated with a bioresorbable scaffold at any time prior to index procedure
4. Cannot provide written informed consent
5. Under judicial protection, tutorship or curatorship
6. Unable to understand and follow study-related instructions or unable to comply with study protocol
7. Active bleeding requiring medical attention (BARC≥2) on randomization visit
8. Life expectancy less than one year
9. Known hypersensitivity or allergy for aspirin, clopidogrel, ticagrelor, prasugrel, cobalt chromium or sirolimus
10. Any planned and anticipated PCI
11. Participation in another trial
12. Pregnant or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4579 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Net adverse clinical endpoints (NACE) defined as a composite of all-cause death, myocardial infarction, stroke and bleeding events defined as BARC 3 or 5 | 11 months
Major adverse cardiac and cerebral events (MACCE) defined as a composite of all-cause death, myocardial infarction and stroke | 11 months
Major or clinically relevant non-major bleeding (MCB) defined as a composite of type 2, 3 and 5 BARC bleeding events | 11 months

SECONDARY OUTCOMES:
All cause death | 14 months
Death from cardiovascular causes | 14 months
Myocardial infarction | 14 months
Stroke | 14 months
Bleeding events | 14 months
Definite or probable stent thrombosis | 14 months
Any target vessel revascularization | 14 months
Urgent target vessel revascularization | 14 months
Urgent non-target vessel revascularization | 14 months
Clinically indicated non-target vessel revascularization | 14 months
Transfusion rates both in patients with and/or without clinically detected over bleeding | 14 months

CONTACTS AND LOCATIONS:
Overall Officials: M. Valgimigli, Prof., Principal Investigator — Cardiocentro Ticino Foundation, Lugano, Switzerland; P. Smits, Dr., Principal Investigator — Maasstad Ziekenhuis Rotterdam, The Netherlands; E. Spitzer, Dr., Study Director — ECRI bv
Locations (138):
- Argentina (2):
  - Buenos Aires Research center, Buenos Aires
  - Interventional Cardiology Sanatorio, Buenos Aires
- Australia (5):
  - The Prince Charles Hospital, Chermside
  - St Vincents Hospital Melbourne, Melbourne
  - Research Center Perth, Perth
  - Research Center Sydney, Sydney
  - Wollongong Research Center, Wollongong
- Austria (2):
  - Research Center , 043-02, Vienna
  - Research Center, 043-01, Vienna
- Research Centre Manama, Manama, Bahrain
- Dhaka Research Center, Dhaka, Bangladesh
- Belgium (6):
  - Research Center Aalst, Aalst
  - Research Center Bonheiden, Bonheiden
  - CHU st.Pierre, Brussels
  - Research Centre Charleroi, Charleroi
  - Research Center Hasselt, Hasselt
  - Research Centre Liège, Liège
- Bulgaria (4):
  - MHAT Sveta Karidad Plovdiv, Plovdiv
  - Sofia Resaerch Center, 359-02, Sofia
  - Sofia Research Center, 359-01, Sofia
  - Sofia Research Center, 359-03, Sofia
- Czechia (2):
  - Research Center Brno, Brno
  - Research Center Phraha, Prague
- Research Center Roskilde, Roskilde, Denmark
- Research Center Tallinn, Tallinn, Estonia
- France (16):
  - Research Center Annecy, Annecy
  - Hospital Prive Saint Martin, Caen
  - Research Centre Caen, Caen
  - Research Centre Créteil, Créteil
  - Research Center Dijon, Dijon
  - Hopital de la Timone, Marseille
  - Research Center Massy, Massy
  - Hospital de Mercy, Metz
  - Research Center Montauban, Montauban
  - Research Centre Montpellier, Montpellier
  - Research Center Nantes, Nantes
  - CHU Nimes, Nîmes
  - Research Center Paris, 033-05, Paris
  - Research Center Paris, 033-06, Paris
  - Research Centre Rouen, Rouen
  - Research Center Saint-Denis, Saint-Denis
- Germany (2):
  - Saarland University, Homburg
  - Cardiology Clinic, Landshut
- Hungary (2):
  - Research Centre Budapest, Budapest
  - Research Center Szeged, Szeged
- India (4):
  - Research Center Chennai, 091-01, Chennai
  - Research Center Chennai, 091-05, Chennai
  - Research Center Coimbatore, Coimbatore
  - Research Center Surat, Sūrat
- Israel (4):
  - Research Center Haifa, Haifa
  - Research Center Jerusalem, Jerusalem
  - Rabin MC, Petah Tikva
  - Research Center Safed, Safed
- Italy (16):
  - Ospedale Lorenzo Bonomo, Andria
  - Azienda Ospedaliera Brotzu, Cagliari
  - Second university of Naples Monaldi Hospital, Caserta
  - Research Center Catania, Catania
  - AOU Policlinico Gaetano Martino, Messina
  - Niguarda, Milan
  - Research Center Milan, 039-01, Milan
  - Research Center Milan, 039-04, Milan
  - Research Center Milan, 039-11, Milan
  - San Donato Hospital, Milan
  - Ospedale Sandro Pertini, Roma
  - Policlinico Casilino, Rome
  - Policlinico Umberto I, Rome
  - Research Center Rozzano, Rozzano
  - Clinic Cardiology, Treviglio
  - Research Center Vimercate, Vimercate
- Japan (11):
  - Kokura Memorial Hospital, Fukuoka
  - Research Center Gifu, Gifu
  - Ichinomiya Municipal Hospital, Ichinomiya
  - St.Marianna University School of Medicine, Kawasaki
  - Aichi Medical University Hospital, Nagakute
  - Japan Red Cross Nagoya Daiichi Hospital (1st), Nagoya
  - Japan Red Cross Nagoya Daini Hospital (2nd), Nagoya
  - Nagoya University Hospital, Nagoya
  - Osaka police Hospital, Osaka
  - St.Luke's International Hospital, Tokyo
  - Research Center Toyoake, Toyoake
- Netherlands (11):
  - Research Center Den Bosch, 's-Hertogenbosch
  - Research Centre Arnhem, Arnhem
  - Research Center Breda, Breda
  - Research Centre Dordrecht, Dordrecht
  - Research Centre Eindhoven, Eindhoven
  - Research Center Emmen, Emmen
  - Research Centre Enschede, Enschede
  - Antonius ziekenhuis, Nieuwegein
  - Research Center Rotterdam, Rotterdam
  - Research Centre Terneuzen, Terneuzen
  - Haga Hospital, The Hague
- Research Center Skopje, Skopje, North Macedonia
- Poland (5):
  - Research Center Krakow, Krakow
  - University Hospital Krakow, Krakow
  - Miedziowe Centrum Zdrowia SA, Lubin
  - Research Center Poznan, Poznan
  - Research Centre Wroclaw, Wroclaw
- Saudi Arabia (2):
  - Research Center Jeddah, Jeddah
  - Research Center Riyadh, Riyadh
- Serbia (3):
  - Researcg Center Belgrade, 381-02, Belgrade
  - Research Center of Serbia, 381-01, Belgrade
  - Research Center Sremska Kamenica, Kamenitz
- Singapore (2):
  - Singapore Research Center, Singapore
  - Tan Tock Seng Hospital, Singapore
- Ljubljana Research Center, Ljubljana, Slovenia
- Research Center Seoul, Seoul, South Korea
- Spain (10):
  - Research Center Alicante, Alicante
  - Research Center Barcelona, 034-07, Barcelona
  - Research Center Barcelona, 034-09, Barcelona
  - Universitario Virgen de la Arrixaca, El Palmar
  - Research Center Huelva, Huelva
  - Hospital Universitario Puerta de hierro, Madrid
  - Research Center Madrid, 034-06, Madrid
  - Research Center Madrid, 034-10, Madrid
  - Hospital Universitario Valdecilla, Santander
  - Research Center Vigo, Vigo
- Sweden (2):
  - Research Center Gavle, Gävle
  - Research Center Orebro, Örebro
- Switzerland (7):
  - Lindenhofspital, Bern
  - Research Centre Bern, Bern
  - Research Centre Fribourg, Fribourg
  - University Hospital Geneva, Geneva
  - Research Centre Liestal, Liestal
  - Research Centre Lugano, Lugano
  - Research Centre Zürich, Zurich
- United Kingdom (12):
  - Research Center Blackburn, Blackburn
  - Research Center Bournemouth, Bournemouth
  - Research Centre Brighton, Brighton
  - Bristol Heart Institute, Bristol
  - St George's Hospital, London
  - Altnagelvin Hospital, Londonderry
  - Manchester Research Center, Manchester
  - Research Center Newcastle, Newcastle upon Tyne
  - Research Center Stevenage, Stevenage
  - Research Centre Stoke-on-Trent, Stoke-on-Trent
  - Research Centre Wolverhampton, Wolverhampton
  - Research Centre Worcester, Worcester
- Vietnam National Heart Institute, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Authors/Task Force members; Windecker S, Kolh P, Alfonso F, Collet JP, Cremer J, Falk V, Filippatos G, Hamm C, Head SJ, Juni P, Kappetein AP, Kastrati A, Knuuti J, Landmesser U, Laufer G, Neumann FJ, Richter DJ, Schauerte P, Sousa Uva M, Stefanini GG, Taggart DP, Torracca L, Valgimigli M, Wijns W, Witkowski A. 2014 ESC/EACTS Guidelines on myocardial revascularization: The Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS)Developed with the special contribution of the European Association of Percutaneous Cardiovascular Interventions (EAPCI). Eur Heart J. 2014 Oct 1;35(37):2541-619. doi: 10.1093/eurheartj/ehu278. Epub 2014 Aug 29. No abstract available. PMID 25173339
- [Background] Roffi M, Patrono C, Collet JP, Mueller C, Valgimigli M, Andreotti F, Bax JJ, Borger MA, Brotons C, Chew DP, Gencer B, Hasenfuss G, Kjeldsen K, Lancellotti P, Landmesser U, Mehilli J, Mukherjee D, Storey RF, Windecker S; ESC Scientific Document Group. 2015 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation: Task Force for the Management of Acute Coronary Syndromes in Patients Presenting without Persistent ST-Segment Elevation of the European Society of Cardiology (ESC). Eur Heart J. 2016 Jan 14;37(3):267-315. doi: 10.1093/eurheartj/ehv320. Epub 2015 Aug 29. No abstract available. PMID 26320110
- [Background] Levine GN, Bates ER, Bittl JA, Brindis RG, Fihn SD, Fleisher LA, Granger CB, Lange RA, Mack MJ, Mauri L, Mehran R, Mukherjee D, Newby LK, O'Gara PT, Sabatine MS, Smith PK, Smith SC, Jr. 2016 ACC/AHA Guideline Focused Update on Duration of Dual Antiplatelet Therapy in Patients With Coronary Artery Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines: An Update of the 2011 ACCF/AHA/SCAI Guideline for Percutaneous Coronary Intervention, 2011 ACCF/AHA Guideline for Coronary Artery Bypass Graft Surgery, 2012 ACC/AHA/ACP/AATS/PCNA/SCAI/STS Guideline for the Diagnosis and Management of Patients With Stable Ischemic Heart Disease, 2013 ACCF/AHA Guideline for the Management of ST-Elevation Myocardial Infarction, 2014 AHA/ACC Guideline for the Management of Patients With Non-ST-Elevation Acute Coronary Syndromes, and 2014 ACC/AHA Guideline on Perioperative Cardiovascular Evaluation and Management of Patients Undergoing Noncardiac Surgery. Circulation 2016
- [Derived] Landi A, Mahfoud F, Frigoli E, Chalkou K, Heg D, Abhaichand RK, Abhyankar AD, Barbato E, Beygui F, Danse PW, Garachemani A, Del Blanco BG, Huber K, Koning R, Kukreja N, Piot C, Quang NN, Tirouvanziam A, Valla M, Smits PC, Valgimigli M, Master Dapt Investigators OBOT. Abbreviated or standard antiplatelet therapy after PCI in HBR patients with chronic kidney disease: a prespecified analysis from the MASTER DAPT trial. EuroIntervention. 2025 Dec 1;21(23):e1445-e1455. doi: 10.4244/EIJ-D-25-00566. PMID 41342080
- [Derived] Bongiovanni D, Landi A, Frigoli E, Heg D, Chalkou K, Bartunek J, Delorme L, Dewilde W, Hildick-Smith D, Leibundgut G, Leonardi S, Lesiak M, Kala P, Kedev S, Roffi M, Stankovic G, Tonino PAL, Velchev V, Vranckx P, Windecker S, Smits PC, Valgimigli M; MASTER DAPT Investigators. Recurrent Events Analysis of MASTER DAPT: Total Ischemic and Bleeding Events After Abbreviated vs Prolonged DAPT in HBR Patients. J Am Coll Cardiol. 2025 Aug 19;86(7):485-498. doi: 10.1016/j.jacc.2025.05.010. Epub 2025 May 22. PMID 40406944
- [Derived] Roffi M, Landi A, Heg D, Frigoli E, Chalkou K, Chevalier B, Ijsselmuiden AJJ, Kastberg R, Komiyama N, Morice MC, Onuma Y, Ozaki Y, Peace A, Pyxaras S, Sganzerla P, Williams R, Xaplanteris P, Vranckx P, Windecker S, Smits PC, Valgimigli M; MASTER DAPT Investigators. Abbreviated or Standard Antiplatelet Therapy After PCI in Diabetic Patients at High Bleeding Risk. JACC Cardiovasc Interv. 2024 Nov 25;17(22):2664-2677. doi: 10.1016/j.jcin.2024.08.030. PMID 39603779
- [Derived] Landi A, Alasnag M, Heg D, Frigoli E, Malik FTN, Gomez-Blazquez I, Pourbaix S, Chieffo A, Spaulding C, Sainz F, Routledge H, Ando G, Testa L, Sciahbasi A, Contractor H, Jepson N, Mieres J, Imran SS, Noor H, Smits PC, Valgimigli M; MASTER DAPT Investigators. Abbreviated or Standard Dual Antiplatelet Therapy by Sex in Patients at High Bleeding Risk: A Prespecified Secondary Analysis of a Randomized Clinical Trial. JAMA Cardiol. 2024 Jan 1;9(1):35-44. doi: 10.1001/jamacardio.2023.4316. PMID 37991745
- [Derived] Landi A, Heg D, Frigoli E, Vranckx P, Windecker S, Siegrist P, Cayla G, Wlodarczak A, Cook S, Gomez-Blazquez I, Feld Y, Seung-Jung P, Mates M, Lotan C, Gunasekaran S, Nanasato M, Das R, Kelbaek H, Teiger E, Escaned J, Ishibashi Y, Montalescot G, Matsuo H, Debeljacki D, Smits PC, Valgimigli M; MASTER DAPT Investigators. Abbreviated or Standard Antiplatelet Therapy in HBR Patients: Final 15-Month Results of the MASTER-DAPT Trial. JACC Cardiovasc Interv. 2023 Apr 10;16(7):798-812. doi: 10.1016/j.jcin.2023.01.366. PMID 37045500
- [Derived] Smits PC, Frigoli E, Vranckx P, Ozaki Y, Morice MC, Chevalier B, Onuma Y, Windecker S, Tonino PAL, Roffi M, Lesiak M, Mahfoud F, Bartunek J, Hildick-Smith D, Colombo A, Stankovic G, Iniguez A, Schultz C, Kornowski R, Ong PJL, Alasnag M, Rodriguez AE, Paradies V, Kala P, Kedev S, Al Mafragi A, Dewilde W, Heg D, Valgimigli M; MASTER DAPT Investigators. Abbreviated Antiplatelet Therapy After Coronary Stenting in Patients With Myocardial Infarction at High Bleeding Risk. J Am Coll Cardiol. 2022 Sep 27;80(13):1220-1237. doi: 10.1016/j.jacc.2022.07.016. PMID 36137672
- [Derived] Valgimigli M, Frigoli E, Vranckx P, Ozaki Y, Morice MC, Chevalier B, Onuma Y, Windecker S, Delorme L, Kala P, Kedev S, Abhaichand RK, Velchev V, Dewilde W, Podolec J, Leibundgut G, Topic D, Schultz C, Stankovic G, Lee A, Johnson T, Tonino PAL, Klotzka A, Lesiak M, Lopes RD, Smits PC, Heg D; MASTER DAPT Investigators. Impact of Medication Nonadherence in a Clinical Trial of Dual Antiplatelet Therapy. J Am Coll Cardiol. 2022 Aug 23;80(8):766-778. doi: 10.1016/j.jacc.2022.04.065. PMID 35981821
- [Derived] Valgimigli M, Smits PC, Frigoli E, Bongiovanni D, Tijssen J, Hovasse T, Mafragi A, Ruifrok WT, Karageorgiev D, Aminian A, Garducci S, Merkely B, Routledge H, Ando K, Diaz Fernandez JF, Cuisset T, Nesa Malik FT, Halabi M, Belle L, Din J, Beygui F, Abhyankar A, Reczuch K, Pedrazzini G, Heg D, Vranckx P; MASTER DAPT Investigators. Duration of antiplatelet therapy after complex percutaneous coronary intervention in patients at high bleeding risk: a MASTER DAPT trial sub-analysis. Eur Heart J. 2022 Sep 1;43(33):3100-3114. doi: 10.1093/eurheartj/ehac284. PMID 35580836
- [Derived] Smits PC, Frigoli E, Tijssen J, Juni P, Vranckx P, Ozaki Y, Morice MC, Chevalier B, Onuma Y, Windecker S, Tonino PAL, Roffi M, Lesiak M, Mahfoud F, Bartunek J, Hildick-Smith D, Colombo A, Stankovic G, Iniguez A, Schultz C, Kornowski R, Ong PJL, Alasnag M, Rodriguez AE, Moschovitis A, Laanmets P, Heg D, Valgimigli M; MASTER DAPT Investigators. Abbreviated Antiplatelet Therapy in Patients at High Bleeding Risk With or Without Oral Anticoagulant Therapy After Coronary Stenting: An Open-Label, Randomized, Controlled Trial. Circulation. 2021 Oct 12;144(15):1196-1211. doi: 10.1161/CIRCULATIONAHA.121.056680. Epub 2021 Aug 29. PMID 34455849
- [Derived] Valgimigli M, Frigoli E, Heg D, Tijssen J, Juni P, Vranckx P, Ozaki Y, Morice MC, Chevalier B, Onuma Y, Windecker S, Tonino PAL, Roffi M, Lesiak M, Mahfoud F, Bartunek J, Hildick-Smith D, Colombo A, Stankovic G, Iniguez A, Schultz C, Kornowski R, Ong PJL, Alasnag M, Rodriguez AE, Moschovitis A, Laanmets P, Donahue M, Leonardi S, Smits PC; MASTER DAPT Investigators. Dual Antiplatelet Therapy after PCI in Patients at High Bleeding Risk. N Engl J Med. 2021 Oct 28;385(18):1643-1655. doi: 10.1056/NEJMoa2108749. Epub 2021 Aug 28. PMID 34449185
- [Derived] Vlieger S, Danzi GB, Kauer F, Oemrawsingh RM, Stojkovic S, IJsselmuiden AJJ, Routledge H, Laanmets P, Roffi M, Frobert O, Baello P, Wlodarczak A, Puentes A, Polad J, Hildick-Smith D. One-year performance of thin-strut cobalt chromium sirolimus-eluting stent versus thicker strut stainless steel biolimus-eluting coronary stent: a propensity-matched analysis of two international all-comers registries. Coron Artery Dis. 2021 Aug 1;32(5):391-396. doi: 10.1097/MCA.0000000000000958. PMID 33060529
- [Derived] Frigoli E, Smits P, Vranckx P, Ozaki Y, Tijssen J, Juni P, Morice MC, Onuma Y, Windecker S, Frenk A, Spaulding C, Chevalier B, Barbato E, Tonino P, Hildick-Smith D, Roffi M, Kornowski R, Schultz C, Lesiak M, Iniguez A, Colombo A, Alasnag M, Mullasari A, James S, Stankovic G, Ong PJL, Rodriguez AE, Mahfoud F, Bartunek J, Moschovitis A, Laanmets P, Leonardi S, Heg D, Sunnaker M, Valgimigli M. Design and rationale of the Management of High Bleeding Risk Patients Post Bioresorbable Polymer Coated Stent Implantation With an Abbreviated Versus Standard DAPT Regimen (MASTER DAPT) Study. Am Heart J. 2019 Mar;209:97-105. doi: 10.1016/j.ahj.2018.10.009. Epub 2018 Nov 22. PMID 30703644